CLINICAL TRIAL: NCT00056628
Title: Study to Evaluate the Effect of Flow-Regulated Ventriculoperitoneal Shunting on Progression of Alzheimer's Disease: An Investigation of the Safety and Effectiveness of the COGNIShunt® CNS Shunt System
Brief Title: COGNIShunt® System for Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunoe (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IA0040; Eunoe protocol ID 2000-01; IDE G970117
Record Dates: First submitted 2003-03-19; First posted 2003-03-20 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2004-10

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Dementia; Ventriculoperitoneal shunt; Tau; ABeta
MeSH Terms: conditions — Alzheimer Disease; Dementia; Pick Disease of the Brain

INTERVENTIONS:
Device: The COGNIShunt® System

SUMMARY:
This is a study of the effect on the progression of Alzheimer's Disease of a surgically implanted shunt (tube) to increase the flow of cerebrospinal fluid and improve the clearance of potential neurotoxins from the fluid bathing the brain.

DETAILED DESCRIPTION:
Cerebrospinal fluid (CSF) is the protective fluid that fills the empty spaces around the brain and spinal cord. CSF is naturally produced and absorbed, but with age abnormal metabolism and clearance of amyloid beta proteins can lead to accumulation of these proteins, resulting in plaque formation, a leading contributor to the progression of Alzheimer's disease (AD). The shunt treatment is designed to drain CSF with these toxic elements from the skull and allow replenishment of normal CSF. This clinical study is designed to determine if this device will stop or slow the progression of Alzheimer's disease.

The COGNIShunt® System is a proprietary device designed to increase the flow of cerebrospinal fluid (CSF) and improve clearance of putative neurotoxins from the CSF that are believed to contribute to the progression of Alzheimer's disease symptoms. This clinical study is designed to determine if this device will stop or slow the progression of Alzheimer's disease. The pivotal study is a prospective, randomized double-blinded, placebo-controlled trial to evaluate the effect of flow-regulated ventriculoperitoneal CSF drainage with the COGNIShunt® system on cognitive and clinical function in approximately 250 participants with Alzheimer's Disease (NINDS/ADRDA criteria). Study participants will be permitted to continue anti-dementia drug therapy if their drug regime has been stable for 3 months prior to entry. This is a two-part study. In Part I, participants will be randomized to receive either a functioning COGNIShunt® System (test/intervention group) or an occluded shunt (control/placebo group). The duration of Part I is nine months, to be followed by an extension phase of an additional 9 months, constituting Part II. During Part II, subjects with occluded shunts have the opportunity to receive a functioning COGNIShunt®, so that all study participants may have open devices during Part II. The total duration of the study is 18 months. Visits to the site include: for screening and baseline (may be done in one or two visits); surgery; and a visit the 1st, 3rd, 6th, 9th, 12th, 15th, and 18th month after surgery.

ELIGIBILITY:
* Participants must meet National Institute of Neurological Disorders and Strokes, and Alzheimer's Disease and Related Disorders Association (NINDS/ADRDA) criteria of probable Alzheimer's disease of mild to moderate severity.
* Age at inclusion into study is between 62 and 85 years. Age at onset of symptoms of Alzheimer's disease must be between 60 and 85 years of age.
* Participants must have no systemic or other brain diseases that could explain deficits in memory or cognition.
* Imaging studies must be consistent with a diagnosis of Alzheimer's disease.
* Hachinski Ischemic Rating Scale score of 4 or less.
* Participants must have sufficient visual and auditory acuity and verbal communication skills to read and hear the testing materials and respond to questions.
* Participants must be able to read and speak English.
* Participants must have a responsible caregiver/informant willing to participate in the study.
* Use of anti-dementia drugs is permitted if participants have been on a stable dose for at least 3 months prior to enrollment.

Exclusion Criteria:

* Family history of early onset Alzheimer's disease.
* History of recent acute myocardial infarction.
* Unstable angina.
* Participants receiving anticoagulants or anti-platelet agents.
* History of malignancy, active systemic infections, clinically significant respiratory dysfunction and/or liver disease.
* History of bleeding disorders, uncontrolled diabetes mellitus and/or hypothyroidism.
* History of stroke.
* Diagnosis of Normal Pressure Hydrocephalus.
* Chronic renal insufficiency.
* History of severe head injury.
* History of alcohol and/or drug abuse.
* Positive FTA, low serum B12.
* Participants exhibiting Parkinsonian signs.

Ages: 62 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2001-01; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Dawn McGuire, MD, Chief Scientific Officer, Study Director — Eunoe, Inc. 643 Bair Island Road, Redwood City, CA 94063

REFERENCES:
- [Background] Silverberg GD, Levinthal E, Sullivan EV, Bloch DA, Chang SD, Leverenz J, Flitman S, Winn R, Marciano F, Saul T, Huhn S, Mayo M, McGuire D. Assessment of low-flow CSF drainage as a treatment for AD: results of a randomized pilot study. Neurology. 2002 Oct 22;59(8):1139-45. doi: 10.1212/01.wnl.0000031794.42077.a1. PMID 12391340
- [Background] Rubenstein E. Relationship of senescence of cerebrospinal fluid circulatory system to dementias of the aged. Lancet. 1998 Jan 24;351(9098):283-5. doi: 10.1016/S0140-6736(97)09234-9. PMID 9457114
- [Background] Silverberg GD, Heit G, Huhn S, Jaffe RA, Chang SD, Bronte-Stewart H, Rubenstein E, Possin K, Saul TA. The cerebrospinal fluid production rate is reduced in dementia of the Alzheimer's type. Neurology. 2001 Nov 27;57(10):1763-6. doi: 10.1212/wnl.57.10.1763. PMID 11723260